CLINICAL TRIAL: NCT03836729
Title: An Open-Label One-way Interaction Clinical Trial to Evaluate the Pharmacokinetic Interactions Between GSK3640254 and Tenofovir Alafenamide/Emtricitabine in Healthy Subjects
Brief Title: Study to Evaluate the Effect of GSK3640254 on the Pharmacokinetics of Tenofovir Alafenamide/Emtricitabine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 208134
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: HIV Infections
Keywords: Human immunodeficiency virus; Sequential; Tenofovir alafenamide; Emtricitabine; GSK3640254
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — emtricitabine tenofovir alafenamide; GSK3640254

STUDY DESIGN:
Intervention Model Description: This is a fixed-sequence 2-period, one-way drug interaction study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAF/FTC followed by TAF/FTC + GSK3640254 (Experimental): Subjects will receive TAF/FTC 25/200 mg QD on Days 1 through 14 in Treatment Period 1. Subjects will be co-administered TAF/FTC 25/200 mg QD with GSK3640254 200 mg QD on Days 1 through 7 in Treatment Period 2.
  Interventions: Drug: Tenofovir alafenamide/emtricitabine; Drug: GSK3640254

INTERVENTIONS:
Drug: Tenofovir alafenamide/emtricitabine — TAF/FTC will be available as 25/200 milligrams (mg) tablet. Subjects will be administered TAF/FTC 25/200 mg QD via the oral route.
Drug: GSK3640254 — GSK3640254 will be available as 100 mg capsule. Subjects will be administered GSK3640254 200 mg capsule QD via the oral route.

SUMMARY:
Human immunodeficiency virus (HIV) infection frequently involves combination drug therapy for its treatment; hence, it is important to understand their interactions and resulting changes in exposure which are associated with medications. This is a Phase-1, open-label, fixed-sequence 2-period, one-way drug interaction study to assess the pharmacokinetic (PK), safety, and tolerability of GSK3640254 and Tenofovir alafenamide/emtricitabine (TAF/FTC) when administered alone and in combination in healthy subjects. The study will consist of a screening period of 28 days before the first dose of study intervention followed by 2 sequential treatment periods. Subjects will be administered TAF/FTC 25/200 milligram (mg) once daily (QD) on Days 1 to 14 of Period 1 followed by co-administration of TAF/FTC 25/200 mg QD with GSK3640254 200 mg QD on Days 1 to 7 of Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Subjects who are healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and ECG).
* Body weight >=50.0 kilograms (kg) (110 pound [lbs]) for men and >=45.0 kilograms [kg] (99 lbs) for women and body mass index (BMI) within the range 18.5 to 31.0 kilograms per meter square (kg/m^2) (inclusive).
* Male or female; A female subject is eligible to participate if she is not pregnant, not breastfeeding and not a woman of childbearing potential (WOCBP).
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A pre-existing condition interfering with normal gastrointestinal (GI) anatomy or motility (e.g.,gastroesophageal reflux disease, gastric ulcers, gastritis), hepatic and/or renal function, that could interfere with the absorption, metabolism and/or excretion of the study drugs or render the subject unable to take oral study intervention.
* Any history of significant underlying psychiatric disorder including, but not limited to, schizophrenia, bipolar disorder with or without psychotic symptoms, other psychotic disorders, or schizotypal (personality) disorder.
* Any history of major depressive disorder with or without suicidal features or anxiety disorders, that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment. Subjects with other conditions such as adjustment disorder or dysthymia that have required shorter term medical therapy (<6 months) without inpatient treatment and are currently well-controlled clinically or resolved may be considered for entry after discussion and agreement with the ViiV Medical Monitor.
* Any pre-existing physical or other psychiatric condition (including alcohol or drug abuse), which, in the opinion of the investigator (with or without psychiatric evaluation), could interfere with the subject's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the subject.
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome.
* History of any kidney disease or current or chronic history of impaired renal function as indicated by an estimated creatinine clearance <80 milliliters per minute (mL/min). Creatinine clearance (CrCL) is estimated by either of the following methods: (a) The Modification of Diet in Renal Disease (MDRD) equation: estimated glomerular filtration rate (eGFR) (milliliter [mL]/minute [min]/1.73 meter square [m^2]) = 175 x (SCr)^-1.154 x (Age)^-0.203 x 0.742 [if female] x 1.212 [if African American] glomerular filtration rate (GFR) is expressed in mL/min/1.73 m^2, SCr is serum creatinine expressed in milligrams per deciliter (mg/dL), and age is expressed in years. (b)The Cockcroft-Gault equation: CrCL(mL/min) ={((l40-age) x weight)/(72xSCr)}x 0.85 (if female) CrCL is expressed in mL/min, age is expressed in years, weight is expressed in kg, and SCr is serum creatinine expressed in mg/dL.
* Presence of Hepatitis B surface antigen (HBsAg) at Screening or within 3 months prior to starting study intervention.
* Positive Hepatitis C antibody test result at Screening or within 3 months prior to starting study intervention AND positive on reflex to Hepatitis C ribonucleic acid (RNA).
* Positive HIV-1 and -2 antigen/antibody immunoassay at Screening.
* ALT >1.5 × upper limit of normal (ULN). A single repeat of ALT is allowed within a single screening period to determine eligibility.
* Bilirubin >1.5 × ULN (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Any acute laboratory abnormality at Screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
* Any Grade 2 to 4 laboratory abnormality at Screening, with the exception of creatine phosphokinase (CPK) and lipid abnormalities (e.g., total cholesterol, triglycerides, etc), and ALT (described above), will exclude a subject from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor. A single repeat of any laboratory abnormality is allowed within a single screening period to determine eligibility.
* A positive test result for drugs of abuse (including marijuana), alcohol, or cotinine (indicating active current smoking) at Screening or before the first dose of study intervention.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and for the duration of the study.
* Treatment with any vaccine within 30 days prior to receiving study intervention.
* Unwillingness to abstain from excessive consumption of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos or their fruit juices within 7 days prior to the first dose of study intervention(s) until the end of the study.
* Participation in another concurrent clinical study or prior clinical study (with the exception of imaging trials) prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the study intervention (whichever is longer).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* Any positive (abnormal) response confirmed by the investigator on a screening clinician- or qualified designee-administered Columbia-Suicide Severity Rating Scale (C-SSRS).
* Any significant arrhythmia or ECG finding (e.g., prior myocardial infarction, sinoatrial pauses, bundle branch block, or conduction abnormality) which, in the opinion of the investigator or VH/GSK Medical Monitor, will interfere with the safety for the individual subject.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate for male: <45 or >100 beats per minute (bpm) and for females: <50 or >100 bpm; PR interval: <120 or >200 milliseconds (msec); QRS duration: <70 or >110 msec and QTcF interval for male: >450 msec and for female: >470 msec. A heart rate from 100 to 110 bpm can be rechecked by ECG or vital signs within 30 minutes to verify eligibility.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 units. One unit is equivalent to 8 grams of alcohol: a half-pint (equivalent to 240 mL) of beer, 1 glass (125 mL) of wine, or 1 (25 mL) measure of spirits.
* Regular use of tobacco- or nicotine-containing products within 3 months prior to Screening.
* History of sensitivity to any of the study medications or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Pene Dumitrescu T, Joshi SR, Xu J, Zhan J, Johnson M, Butcher L, Zimmerman E, Webster L, Davidson AM, Lataillade M, Min S. A Phase I Evaluation of the Pharmacokinetics and Tolerability of the HIV-1 Maturation Inhibitor GSK3640254 and Tenofovir Alafenamide/Emtricitabine in Healthy Participants. Antimicrob Agents Chemother. 2021 May 18;65(6):e02173-20. doi: 10.1128/AAC.02173-20. Print 2021 May 18. PMID 33753329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, single-sequence one-way interaction drug interaction study to investigate the effect of GSK3640254 on the pharmacokinetics (PK) of tenofovir alafenamide (TAF) and emtricitabine (FTC).
Pre-assignment Details: A total of 16 participants were enrolled in the study.
Groups:
- TAF/FTC Followed by TAF/FTC+GSK3640254: Participants in Period 1 received 25 milligram (mg) of TAF and 200 mg of FTC once daily (QD) on Days 1 through 14. In Period 2 participant's co-administered 25 mg TAF and 200 mg FTC QD along with GSK3640254 200 mg QD on Days 1 through 7. There was no washout period between two periods.
Period: Treatment Period 1 (Up to Day 14)
Arm/Group | TAF/FTC Followed by TAF/FTC+GSK3640254
Started | 16
Completed | 16
Not Completed | 0
Period: Treatment Period 2 (Up to Day 7)
Arm/Group | TAF/FTC Followed by TAF/FTC+GSK3640254
Started | 16
Completed | 15
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- TAF/FTC Followed by TAF/FTC+GSK3640254: Participants in Period 1 received 25 mg of TAF and 200 mg of FTC QD on Days 1 through 14. In Period 2 participant's co-administered 25 mg TAF and 200 mg FTC QD along with GSK3640254 200 mg QD on Days 1 through 7. There was no washout period between two periods.
Arm/Group | TAF/FTC Followed by TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.9 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1
  Asian: East Asian Heritage | 1
  Black or African American | 7
  Native Hawaiian or other pacific islander | 1
  White:White/Caucasian/European Heritage | 6

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Area Under the Plasma Concentration-time Curve From Time 0 to the End of the Dosing Interval at Steady State (AUC [0-tau]) of TAF
Description: Blood samples were collected at indicated time-points for analysis of AUC (0-tau). Pharmacokinetic (PK) parameters were calculated by standard non-compartmental analysis. PK Parameter Population included all participants who underwent plasma PK sampling and had evaluable PK parameters estimated.
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 1 Day 14
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- TAF/FTC: Participants in Period 1 received 25 mg of TAF and 200 mg of FTC QD on Days 1 through 14. There was no washout period between two periods.
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Hours*nanogram per milliliter | 250.4 (58.2)

2. Primary Outcome: Period 2: AUC (0-tau) of TAF
Description: Blood samples were collected at indicated time-points for analysis of AUC (0-tau). PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Groups:
- TAF/FTC+GSK3640254: In Period 2 participants co-administered 25 mg TAF and 200 mg FTC QD along with GSK3640254 200 mg QD on Days 1 through 7. There was no washout period between two periods.
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Hours*nanogram per milliliter | 215.4 (36.3)

3. Primary Outcome: Period 1: Maximum Observed Concentration (Cmax) of TAF
Description: Blood samples were collected at indicated time-points for analysis of Cmax. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 1 Day 14
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Nanogram per milliliter | 203.4 (56.1)

4. Primary Outcome: Period 2: Cmax of TAF
Description: as for outcome 3
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Nanogram per milliliter | 175.1 (44.4)

5. Primary Outcome: Period 1: AUC (0-tau) of FTC
Description: as for outcome 2
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 1 Day 14
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Hours*nanogram per milliliter | 9787.5 (15.5)

6. Primary Outcome: Period 2: AUC (0-tau) of FTC
Description: as for outcome 2
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Hours*nanogram per milliliter | 9421.0 (14.4)

7. Primary Outcome: Period 1:Cmax of FTC
Description: as for outcome 3
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 1 Day 14
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Nanogram per milliliter | 1811 (15.9)

8. Primary Outcome: Period 2:Cmax of FTC
Description: as for outcome 3
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Nanogram per milliliter | 1701 (20.9)

9. Primary Outcome: Period 1: Plasma Concentration at the End of the Dosing Interval (Ctau) of FTC
Description: Blood samples were collected at indicated time-points for analysis of Ctau. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 1 Day 14
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Nanogram per milliliter | 71.81 (25.5)

10. Primary Outcome: Period 2: Ctau of FTC
Description: as for outcome 9
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Nanogram per milliliter | 82.92 (29.1)

11. Primary Outcome: Period 1: AUC (0-tau) of Tenofovir (TFV)
Description: as for outcome 2
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 1 Day 14
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Hours*nanogram per milliliter | 221.9 (18.3)

12. Primary Outcome: Period 2: AUC (0-tau) of TFV
Description: as for outcome 2
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Hours*nanogram per milliliter | 229.1 (21.5)

13. Primary Outcome: Period 1: Cmax of TFV
Description: as for outcome 3
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 1 Day 14
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Nanogram per milliliter | 13.14 (17.8)

14. Primary Outcome: Period 2: Cmax of TFV
Description: as for outcome 3
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Nanogram per milliliter | 13.30 (20.8)

15. Primary Outcome: Period 1: Ctau of TFV
Description: as for outcome 9
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 1 Day 14
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Nanogram per milliliter | 7.688 (20.4)

16. Primary Outcome: Period 2: Ctau of TFV
Description: as for outcome 9
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Nanogram per milliliter | 8.244 (22.9)

17. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAE)
Description: An adverse events (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; other important medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before
Time Frame: Up to Day 24
Population: Safety Population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | TAF/FTC | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16 | 15
Participants
  Non-SAEs | 9 | 3
  SAEs | 0 | 0

18. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter of Platelet Count, Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameters like platelet count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, and 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Giga cells per liter
  Basophils, Period 1 Day 7 | -0.005 (0.0167)
  Basophils, Period 1 Day 14 | -0.006 (0.0260)
  Eosinophils, Period 1 Day 7 | -0.021 (0.0795)
  Eosinophils, Period 1 Day 14 | -0.020 (0.1531)
  Monocytes, Period 1 Day 7 | 0.014 (0.1808)
  Monocytes, Period 1 Day 14 | 0.049 (0.2718)
  Leukocytes, Period 1 Day 7 | -0.08 (1.795)
  Leukocytes, Period 1 Day 14 | 0.27 (2.191)
  Lymphocytes, Period 1 Day 7 | -0.246 (0.3089)
  Lymphocytes, Period 1 Day 14 | -0.262 (0.4138)
  Neutrophils, Period 1 Day 7 | 0.188 (1.5473)
  Neutrophils, Period 1 Day 14 | 0.513 (1.7986)
  Platelets, Period 1 Day 7 | 3.3 (21.23)
  Platelets, Period 1 Day 14 | 21.8 (35.37)

19. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter of Platelet Count, Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils
Description: Blood samples were collected at indicated timepoints for analysis for hematology parameters like platelet count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Giga cells per liter
  Basophils, Period 2 Day 3, n= 15: number analyzed (Participants) | 15
  Basophils, Period 2 Day 3, n= 15 | -0.004 (0.0196)
  Basophils, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Basophils, Period 2 Day 7, n= 15 | -0.002 (0.0204)
  Basophils, Period 2 Day 9, n= 15: number analyzed (Participants) | 15
  Basophils, Period 2 Day 9, n= 15 | 0.003 (0.0150)
  Eosinophils, Period 2 Day 3, n=15: number analyzed (Participants) | 15
  Eosinophils, Period 2 Day 3, n=15 | -0.023 (0.0811)
  Eosinophils, Period 2 Day 7, n=15: number analyzed (Participants) | 15
  Eosinophils, Period 2 Day 7, n=15 | -0.039 (0.1058)
  Eosinophils, Period 2 Day 9, n=16 | -0.043 (0.1093)
  Monocytes, Period 2 Day 3, n= 16 | -0.053 (0.1895)
  Monocytes, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Monocytes, Period 2 Day 7, n= 15 | -0.077 (0.1709)
  Monocytes, Period 2 Day 9, n= 15: number analyzed (Participants) | 15
  Monocytes, Period 2 Day 9, n= 15 | -0.104 (0.1672)
  Leukocytes, Period 2 Day 3, n= 16 | -1.06 (1.188)
  Leukocytes, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Leukocytes, Period 2 Day 7, n= 15 | -0.61 (1.050)
  Leukocytes, Period 2 Day 9, n= 15: number analyzed (Participants) | 15
  Leukocytes, Period 2 Day 9, n= 15 | -0.49 (1.193)
  Lymphocytes, Period 2 Day 3, n= 16 | -0.158 (0.2296)
  Lymphocytes, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Lymphocytes, Period 2 Day 7, n= 15 | -0.105 (0.2306)
  Lymphocytes, Period 2 Day 9, n= 15: number analyzed (Participants) | 15
  Lymphocytes, Period 2 Day 9, n= 15 | -0.111 (0.2728)
  Neutrophils, Period 2 Day 3, n= 16 | -0.868 (0.9597)
  Neutrophils, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Neutrophils, Period 2 Day 7, n= 15 | -0.417 (0.9069)
  Neutrophils, Period 2 Day 9, n= 15: number analyzed (Participants) | 15
  Neutrophils, Period 2 Day 9, n= 15 | -0.282 (1.0161)
  Platelets, Period 2 Day 3, n= 16 | 9.2 (20.41)
  Platelets, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Platelets, Period 2 Day 7, n= 15 | 19.8 (43.02)
  Platelets, Period 2 Day 9, n= 15: number analyzed (Participants) | 15
  Platelets, Period 2 Day 9, n= 15 | 16.2 (38.11)

20. Secondary Outcome: Period 1: Absolute Values of the Hematology Parameter of Platelet Count, Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameters like platelet count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, and 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Giga cells per liter
  Basophils, Period 1 Baseline | 0.046 (0.0216)
  Basophils, Period 1 Day 7 | 0.041 (0.0189)
  Basophils, Period 1 Day 14 | 0.040 (0.0256)
  Eosinophils, Period 1 Baseline | 0.225 (0.1918)
  Eosinophils, Period 1 Day 7 | 0.204 (0.1737)
  Eosinophils, Period 1 Day 14 | 0.205 (0.1766)
  Monocytes, Period 1 Baseline | 0.522 (0.1147)
  Monocytes, Period 1 Day 7 | 0.536 (0.2063)
  Monocytes, Period 1 Day 14 | 0.571 (0.2830)
  Leukocytes, Period 1 Baseline | 6.18 (1.336)
  Leukocytes, Period 1 Day 7 | 6.10 (2.024)
  Leukocytes, Period 1 Day 14 | 6.45 (2.231)
  Lymphocytes, Period 1 Baseline | 1.945 (0.7419)
  Lymphocytes, Period 1 Day 7 | 1.699 (0.5822)
  Lymphocytes, Period 1 Day 14 | 1.683 (0.4988)
  Neutrophils, Period 1 Baseline | 3.441 (0.9719)
  Neutrophils, Period 1 Day 7 | 3.628 (1.9503)
  Neutrophils, Period 1 Day 14 | 3.954 (1.9141)
  Platelets, Period 1 Baseline | 253.3 (49.81)
  Platelets, Period 1 Day 7 | 256.6 (49.72)
  Platelets, Period 1 Day 14 | 275.1 (53.39)

21. Secondary Outcome: Period 2: Absolute Values of the Hematology Parameter of Platelet Count, Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameters like platelet count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Giga cells per liter
  Basophils, Period 2 Baseline, n= 16 | 0.040 (0.0256)
  Basophils, Period 2 Day 3, n= 15: number analyzed (Participants) | 15
  Basophils, Period 2 Day 3, n= 15 | 0.036 (0.0182)
  Basophils, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Basophils, Period 2 Day 7, n= 15 | 0.038 (0.0152)
  Basophils, Period 2 Day 9, n= 15: number analyzed (Participants) | 15
  Basophils, Period 2 Day 9, n= 15 | 0.043 (0.0232)
  Eosinophils, Period 2 Baseline, n= 16 | 0.208 (0.1764)
  Eosinophils, Period 2 Day 3, n= 15: number analyzed (Participants) | 15
  Eosinophils, Period 2 Day 3, n= 15 | 0.185 (0.1533)
  Eosinophils, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Eosinophils, Period 2 Day 7, n= 15 | 0.157 (0.1405)
  Eosinophils, Period 2 Day 9, n= 16 | 0.153 (0.1384)
  Monocytes, Period 2 Baseline, n= 16 | 0.545 (0.2127)
  Monocytes, Period 2 Day 3, n= 16 | 0.492 (0.1975)
  Monocytes, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Monocytes, Period 2 Day 7, n= 15 | 0.448 (0.1472)
  Monocytes, Period 2 Day 9, n= 15: number analyzed (Participants) | 15
  Monocytes, Period 2 Day 9, n= 15 | 0.421 (0.1212)
  Leukocytes, Period 2 Baseline, n= 16 | 6.20 (1.752)
  Leukocytes, Period 2 Day 3, n= 16 | 5.14 (1.035)
  Leukocytes, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Leukocytes, Period 2 Day 7, n= 15 | 5.39 (1.311)
  Leukocytes, Period 2 Day 9, n= 15: number analyzed (Participants) | 15
  Leukocytes, Period 2 Day 9, n= 15 | 5.51 (1.415)
  Lymphocytes, Period 2 Baseline, n= 16 | 1.718 (0.4814)
  Lymphocytes, Period 2 Day 3, n= 16 | 1.560 (0.3786)
  Lymphocytes, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Lymphocytes, Period 2 Day 7, n= 15 | 1.570 (0.4116)
  Lymphocytes, Period 2 Day 9, n= 15: number analyzed (Participants) | 15
  Lymphocytes, Period 2 Day 9, n= 15 | 1.563 (0.4236)
  Neutrophils, Period 2 Baseline, n= 16 | 3.724 (1.3787)
  Neutrophils, Period 2 Day 3, n= 16 | 2.857 (0.8106)
  Neutrophils, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Neutrophils, Period 2 Day 7, n= 15 | 3.189 (1.0515)
  Neutrophils, Period 2 Day 9, n= 15: number analyzed (Participants) | 15
  Neutrophils, Period 2 Day 9, n= 15 | 3.324 (1.1988)
  Platelets, Period 2 Baseline, n= 16 | 274.3 (51.10)
  Platelets, Period 2 Day 3, n= 16 | 283.4 (54.62)
  Platelets, Period 2 Day 7, n= 15: number analyzed (Participants) | 15
  Platelets, Period 2 Day 7, n= 15 | 294.0 (54.62)
  Platelets, Period 2 Day 9, n= 15: number analyzed (Participants) | 15
  Platelets, Period 2 Day 9, n= 15 | 290.4 (73.92)

22. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter of Hematocrit
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like hematocrit. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Proportion of red blood cells in blood
  Day 7 | 0.0121 (0.01389)
  Day 14 | 0.0189 (0.01304)

23. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter of Hematocrit
Description: Blood samples were collected at indicated time-points for analysis for hematology parameter like hematocrit. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Groups:
- TAF/FTC+GSK3640254: In Period 2 participant's co-administered 25 mg TAF and 200 mg FTC QD along with GSK3640254 200 mg QD on Days 1 through 7. There was no washout period between two periods.
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Proportion of red blood cells in blood
  Day 3, n= 16 | -0.0147 (0.00982)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | -0.0007 (0.01369)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | -0.0204 (0.01371)

24. Secondary Outcome: Period 1: Absolute Values of the Hematology Parameter: Hematocrit
Description: Blood samples were collected at indicated time points for analysis for hematology parameter like hematocrit. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Proportion of red blood cells in blood
  Baseline | 0.4264 (0.01891)
  Day 7 | 0.4384 (0.02358)
  Day 14 | 0.4453 (0.01997)

25. Secondary Outcome: Period 2: Absolute Values of the Hematology Parameter: Hematocrit
Description: Blood samples were collected at indicated time-points for analysis for hematology parameter like hematocrit. Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Proportion of red blood cells in blood
  Baseline, n= 16 | 0.4453 (0.01997)
  Day 3, n= 16 | 0.4306 (0.01780)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | 0.4444 (0.02234)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | 0.4247 (0.01518)

26. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter of Hemoglobin
Description: Blood samples were collected at indicated timepoints for analysis for hematology parameter like hemoglobin. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Grams per liter
  Day 7 | 6.1 (4.51)
  Day 14 | 8.4 (3.98)

27. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter of Hemoglobin
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like hemoglobin. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Grams per liter
  Day 3, n= 16 | -3.9 (3.51)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | -1.1 (4.58)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | -6.4 (5.55)

28. Secondary Outcome: Period 1: Absolute Values of the Hematology Parameter: Hemoglobin
Description: Blood samples were collected at indicated time-points for analysis for hematology parameter like hemoglobin. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Grams per liter
  Baseline | 142.0 (6.70)
  Day 7 | 148.1 (8.11)
  Day 14 | 150.4 (7.45)

29. Secondary Outcome: Period 2: Absolute Values of the Hematology Parameter: Hemoglobin
Description: Blood samples were collected at indicated time-points for analysis for hematology parameter like hemoglobin. Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Grams per liter
  Baseline, n= 16 | 150.4 (7.45)
  Day 3, n= 16 | 146.4 (6.37)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | 149.1 (7.26)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | 143.9 (5.19)

30. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter of Mean Corpuscle Hemoglobin (MCH)
Description: Blood samples were collected at indicated timepoints for analysis of hematology parameter like MCH. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Picograms
  Day 7 | 0.13 (0.272)
  Day 14 | 0.36 (0.276)

31. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter of MCH
Description: Blood samples were collected at indicated timepoints for analysis for hematology parameter like MCH. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Picograms
  Day 3, n= 16 | -0.11 (0.205)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | -0.21 (0.203)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | -0.17 (0.253)

32. Secondary Outcome: Period 1: Absolute Values of the Hematology Parameter: MCH
Description: Blood samples were collected at indicated time-points for analysis for hematology parameter like MCH. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Picograms
  Baseline | 28.63 (1.780)
  Day 7 | 28.75 (1.687)
  Day 14 | 28.98 (1.690)

33. Secondary Outcome: Period 2: Absolute Values of the Hematology Parameter: MCH
Description: Blood samples were collected at indicated time-points for analysis of hematology parameter like MCH. Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Picograms
  Baseline, n= 16 | 28.98 (1.690)
  Day 3, n= 16 | 28.88 (1.699)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | 28.83 (1.630)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | 28.87 (1.702)

34. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter of Mean Corpuscle Volume (MCV)
Description: Blood samples were collected at indicated time-points for analysis for hematology parameter like MCV. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Femtoliters
  Day 7 | -0.83 (0.620)
  Day 14 | -0.07 (0.712)

35. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter of MCV
Description: Blood samples were collected at indicated timepoints for analysis for hematology parameter like MCV. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Femtoliters
  Day 3, n= 16 | -1.02 (0.483)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | -0.17 (0.472)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | -0.82 (0.499)

36. Secondary Outcome: Period 1: Absolute Values of the Hematology Parameter: MCV
Description: Blood samples were collected at indicated time-points for analysis for hematology parameter like MCV. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Femtoliters
  Baseline | 85.92 (4.690)
  Day 7 | 85.09 (4.504)
  Day 14 | 85.85 (4.492)

37. Secondary Outcome: Period 2: Absolute Values of the Hematology Parameter: MCV
Description: Blood samples were collected at indicated time-points for analysis for hematology parameter like MCV. Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Femtoliters
  Baseline, n= 16 | 85.85 (4.492)
  Day 3, n= 16 | 84.83 (4.490)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | 85.85 (4.491)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | 85.20 (4.601)

38. Secondary Outcome: Period 1: Change From Baseline in Hematology Parameter of Erythrocytes
Description: Blood samples were collected at indicated time-points for analysis for hematology parameter like erythrocytes. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Trillion cells per liter
  Day 7 | 0.189 (0.1485)
  Day 14 | 0.226 (0.1360)

39. Secondary Outcome: Period 2: Change From Baseline in Hematology Parameter of Erythrocytes
Description: Blood samples were collected at indicated time-points for analysis for hematology parameter like erythrocytes. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Trillion cells per liter
  Day 3, n= 16 | -0.113 (0.1123)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | 0.000 (0.1466)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | -0.189 (0.1697)

40. Secondary Outcome: Period 1: Absolute Values of the Hematology Parameter: Erythrocytes
Description: Blood samples were collected at indicated time-points for analysis for hematology parameter like erythrocytes. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Trillion cells per liter
  Baseline | 4.977 (0.3351)
  Day 7 | 5.166 (0.3679)
  Day 14 | 5.203 (0.3604)

41. Secondary Outcome: Period 2: Absolute Values of the Hematology Parameter: Erythrocytes
Description: Blood samples were collected at indicated time-points for analysis for hematology parameter like erythrocytes. Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Trillion cells per liter
  Baseline, n= 16 | 5.203 (0.3604)
  Day 3, n= 16 | 5.090 (0.3395)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | 5.190 (0.4087)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | 5.001 (0.3446)

42. Secondary Outcome: Period 1: Change From Baseline in Clinical Chemistry Parameter of Glucose, Anion Gap, Cholesterol, Calcium, Potassium, Sodium, Blood Urea Nitrogen (BUN), Carbon Dioxide (CO2), Chloride and Phosphorus
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of glucose, calcium, potassium, sodium, BUN, anion gap, CO2, chloride and phosphorus. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Millimoles per Liter
  Glucose, Day 7 | -0.160 (0.3793)
  Glucose, Day 14 | -0.320 (0.3432)
  Cholesterol, Day 7 | -0.004 (0.3735)
  Cholesterol, Day 14 | -0.389 (0.3533)
  Anion gap, Day 7 | 1.9 (2.08)
  Anion gap, Day 14 | 2.2 (1.42)
  Calcium, Day 7 | 0.028 (0.0780)
  Calcium, Day 14 | 0.028 (0.0556)
  CO2, Day 7 | -1.6 (1.93)
  CO2, Day 14 | -0.9 (1.20)
  Chloride, Day 7 | -1.1 (1.06)
  Chloride, Day 14 | -2.0 (1.46)
  Phosphate, Day 7 | 0.017 (0.0960)
  Phosphate, Day 14 | 0.026 (0.1330)
  Potassium, Day 7 | 0.03 (0.304)
  Potassium, Day 14 | -0.03 (0.328)
  Sodium, Day 7 | -0.6 (1.45)
  Sodium, Day 14 | -0.6 (1.59)
  Triglycerides, Day 7 | 0.092 (0.4841)
  Triglycerides, Day 14 | -0.044 (0.4569)
  BUN, Day 7 | -0.018 (1.2157)
  BUN, Day 14 | -0.195 (1.0640)

43. Secondary Outcome: Period 2: Change From Baseline in Clinical Chemistry Parameter of Glucose, Anion Gap, Cholesterol, Calcium, Potassium, Sodium, BUN, CO2, Chloride and Phosphorus
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of glucose, calcium, potassium, sodium, BUN, anion gap, CO2, chloride and phosphorus. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Millimoles per Liter
  Glucose, Day 3, n= 15: number analyzed (Participants) | 15
  Glucose, Day 3, n= 15 | 0.236 (0.2463)
  Glucose, Day 7, n= 15: number analyzed (Participants) | 15
  Glucose, Day 7, n= 15 | 0.315 (0.3282)
  Glucose, Day 9, n= 15: number analyzed (Participants) | 15
  Glucose, Day 9, n= 15 | 0.136 (0.2433)
  Cholesterol, Day 3, n=15: number analyzed (Participants) | 15
  Cholesterol, Day 3, n=15 | 0.011 (0.2372)
  Cholesterol, Day 7, n= 15: number analyzed (Participants) | 15
  Cholesterol, Day 7, n= 15 | 0.102 (0.3899)
  Cholesterol, Day 9, n= 16 | 0.030 (0.4594)
  Anion gap, Day 3, n= 16 | -0.4 (1.82)
  Anion gap, Day 7, n= 15: number analyzed (Participants) | 15
  Anion gap, Day 7, n= 15 | -0.5 (1.73)
  Anion gap, Day 9, n= 15: number analyzed (Participants) | 15
  Anion gap, Day 9, n= 15 | -0.3 (1.67)
  Calcium, Day 3, n= 16 | 0.013 (0.0478)
  Calcium, Day 7, n= 15: number analyzed (Participants) | 15
  Calcium, Day 7, n= 15 | 0.037 (0.0568)
  Calcium, Day 9, n= 15: number analyzed (Participants) | 15
  Calcium, Day 9, n= 15 | 0.033 (0.0628)
  CO2, Day 3, n= 16 | -0.5 (1.26)
  CO2, Day 7, n= 15: number analyzed (Participants) | 15
  CO2, Day 7, n= 15 | -0.1 (1.36)
  CO2, Day 9, n= 15: number analyzed (Participants) | 15
  CO2, Day 9, n= 15 | -0.4 (1.18)
  Chloride, Day 3, n= 16 | 2.3 (1.20)
  Chloride, Day 7, n= 15: number analyzed (Participants) | 15
  Chloride, Day 7, n= 15 | 0.6 (1.35)
  Chloride, Day 9, n= 15: number analyzed (Participants) | 15
  Chloride, Day 9, n= 15 | 1.3 (1.72)
  Phosphate, Day 3, n= 16 | 0.062 (0.0683)
  Phosphate, Day 7, n= 15: number analyzed (Participants) | 15
  Phosphate, Day 7, n= 15 | 0.002 (0.0800)
  Phosphate, Day 9, n= 15: number analyzed (Participants) | 15
  Phosphate, Day 9, n= 15 | 0.007 (0.0584)
  Potassium, Day 3, n= 16 | 0.01 (0.284)
  Potassium, Day 7, n= 15: number analyzed (Participants) | 15
  Potassium, Day 7, n= 15 | -0.03 (0.213)
  Potassium, Day 9, n= 15: number analyzed (Participants) | 15
  Potassium, Day 9, n= 15 | 0.10 (0.344)
  Sodium, Day 3, n= 16 | 1.4 (1.36)
  Sodium, Day 7, n= 15: number analyzed (Participants) | 15
  Sodium, Day 7, n= 15 | 0.1 (1.53)
  Sodium, Day 9, n= 15: number analyzed (Participants) | 15
  Sodium, Day 9, n= 15 | 0.6 (1.06)
  Triglycerides, Day 3, n= 16 | -0.003 (0.1753)
  Triglycerides, Day 7, n= 15: number analyzed (Participants) | 15
  Triglycerides, Day 7, n= 15 | 0.111 (0.2414)
  Triglycerides, Day 9, n= 15: number analyzed (Participants) | 15
  Triglycerides, Day 9, n= 15 | -0.049 (0.2747)
  BUN, Day 3, n= 16 | 0.312 (0.5567)
  BUN, Day 7, n= 15: number analyzed (Participants) | 15
  BUN, Day 7, n= 15 | -0.031 (0.5038)
  BUN, Day 9, n= 15: number analyzed (Participants) | 15
  BUN, Day 9, n= 15 | -0.028 (0.4521)

44. Secondary Outcome: Period 1: Absolute Values of Clinical Chemistry Parameter of Glucose, Anion Gap, Cholesterol, Calcium, Potassium, Sodium, BUN, CO2, Chloride and Phosphorus
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameter of glucose, calcium, potassium, sodium, BUN, anion gap, CO2, chloride and phosphorus. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Millimoles per Liter
  Glucose, Baseline | 5.111 (0.3747)
  Glucose, Day 7 | 4.951 (0.2587)
  Glucose, Day 14 | 4.791 (0.2662)
  Cholesterol, Baseline | 4.253 (0.7938)
  Cholesterol, Day 7 | 4.249 (0.8494)
  Cholesterol, Day 14 | 3.864 (0.6087)
  Anion gap, Baseline | 8.7 (1.08)
  Anion gap, Day 7 | 10.6 (2.25)
  Anion gap, Day 14 | 10.9 (1.45)
  Calcium, Baseline | 2.359 (0.0697)
  Calcium, Day 7 | 2.387 (0.0663)
  Calcium, Day 14 | 2.387 (0.0637)
  CO2, Baseline | 31.7 (1.49)
  CO2, Day 7 | 30.1 (1.86)
  CO2, Day 14 | 30.8 (1.38)
  Chloride, Baseline | 103.3 (1.84)
  Chloride, Day 7 | 102.2 (1.72)
  Chloride, Day 14 | 101.3 (2.32)
  Phosphate, Baseline | 1.078 (0.1301)
  Phosphate, Day 7 | 1.094 (0.1202)
  Phosphate, Day 14 | 1.103 (0.0807)
  Potassium, Baseline | 4.25 (0.225)
  Potassium, Day 7 | 4.28 (0.161)
  Potassium, Day 14 | 4.22 (0.279)
  Sodium, Baseline | 139.4 (1.45)
  Sodium, Day 7 | 138.8 (1.77)
  Sodium, Day 14 | 138.8 (1.69)
  Triglycerides, Baseline | 1.076 (0.5825)
  Triglycerides, Day 7 | 1.168 (0.3759)
  Triglycerides, Day 14 | 1.033 (0.3034)
  BUN, Baseline | 4.441 (1.2792)
  BUN, Day 7 | 4.423 (0.9623)
  BUN, Day 14 | 4.246 (0.7820)

45. Secondary Outcome: Period 2: Absolute Values of Clinical Chemistry Parameter of Glucose, Anion Gap, Cholesterol, Calcium, Potassium, Sodium, BUN, CO2, Chloride and Phosphorus
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of glucose, calcium, potassium, sodium, BUN, anion gap, CO2, chloride and phosphorus. Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Millimoles per Liter
  Glucose, Baseline, n= 16 | 4.791 (0.2662)
  Glucose, Day 3, n= 15: number analyzed (Participants) | 15
  Glucose, Day 3, n= 15 | 5.027 (0.2894)
  Glucose, Day 7, n= 15: number analyzed (Participants) | 15
  Glucose, Day 7, n= 15 | 5.129 (0.3388)
  Glucose, Day 9, n= 15: number analyzed (Participants) | 15
  Glucose, Day 9, n= 15 | 4.950 (0.3360)
  Cholesterol, Baseline, n= 16 | 3.864 (0.6087)
  Cholesterol, Day 3, n=15: number analyzed (Participants) | 15
  Cholesterol, Day 3, n=15 | 3.875 (0.6509)
  Cholesterol, Day 7, n= 15: number analyzed (Participants) | 15
  Cholesterol, Day 7, n= 15 | 3.894 (0.7575)
  Cholesterol, Day 9, n= 16 | 3.822 (0.7838)
  Anion gap, Baseline, n= 16 | 10.9 (1.45)
  Anion gap, Day 3, n= 16 | 10.5 (1.37)
  Anion gap, Day 7, n= 15: number analyzed (Participants) | 15
  Anion gap, Day 7, n= 15 | 10.3 (1.28)
  Anion gap, Day 9, n= 15: number analyzed (Participants) | 15
  Anion gap, Day 9, n= 15 | 10.5 (0.74)
  Calcium, Baseline, n= 16 | 2.387 (0.0637)
  Calcium, Day 3, n= 16 | 2.399 (0.0682)
  Calcium, Day 7, n= 15: number analyzed (Participants) | 15
  Calcium, Day 7, n= 15 | 2.424 (0.0693)
  Calcium, Day 9, n= 15: number analyzed (Participants) | 15
  Calcium, Day 9, n= 15 | 2.421 (0.0670)
  CO2, Baseline, n= 16 | 30.8 (1.38)
  CO2, Day 3, n= 16 | 30.3 (1.96)
  CO2, Day 7, n= 15: number analyzed (Participants) | 15
  CO2, Day 7, n= 15 | 30.7 (1.91)
  CO2, Day 9, n= 15: number analyzed (Participants) | 15
  CO2, Day 9, n= 15 | 30.5 (1.30)
  Chloride, Baseline, n= 16 | 101.3 (2.32)
  Chloride, Day 3, n= 16 | 103.6 (1.50)
  Chloride, Day 7, n= 15: number analyzed (Participants) | 15
  Chloride, Day 7, n= 15 | 101.9 (1.62)
  Chloride, Day 9, n= 15: number analyzed (Participants) | 15
  Chloride, Day 9, n= 15 | 102.7 (1.50)
  Phosphate, Baseline, n= 16 | 1.103 (0.0807)
  Phosphate, Day 3, n= 16 | 1.165 (0.1007)
  Phosphate, Day 7, n= 15: number analyzed (Participants) | 15
  Phosphate, Day 7, n= 15 | 1.112 (0.1097)
  Phosphate, Day 9, n= 15: number analyzed (Participants) | 15
  Phosphate, Day 9, n= 15 | 1.117 (0.0952)
  Potassium, Baseline, n= 16 | 4.22 (0.279)
  Potassium, Day 3, n= 16 | 4.23 (0.241)
  Potassium, Day 7, n= 15: number analyzed (Participants) | 15
  Potassium, Day 7, n= 15 | 4.21 (0.236)
  Potassium, Day 9, n= 15: number analyzed (Participants) | 15
  Potassium, Day 9, n= 15 | 4.35 (0.226)
  Sodium, Baseline, n= 16 | 138.8 (1.69)
  Sodium, Day 3, n= 16 | 140.2 (1.56)
  Sodium, Day 7, n= 15: number analyzed (Participants) | 15
  Sodium, Day 7, n= 15 | 138.8 (1.42)
  Sodium, Day 9, n=15: number analyzed (Participants) | 15
  Sodium, Day 9, n=15 | 139.3 (1.18)
  Triglycerides, Baseline, n= 16 | 1.033 (0.3034)
  Triglycerides, Day 3, n= 16 | 1.029 (0.3440)
  Triglycerides, Day 7, n= 15: number analyzed (Participants) | 15
  Triglycerides, Day 7, n= 15 | 1.120 (0.4358)
  Triglycerides, Day 9, n= 15: number analyzed (Participants) | 15
  Triglycerides, Day 9, n= 15 | 0.961 (0.4320)
  BUN, Baseline, n= 16 | 4.246 (0.7820)
  BUN, Day 3, n= 16 | 4.558 (0.8267)
  BUN, Day 7, n= 15: number analyzed (Participants) | 15
  BUN, Day 7, n= 15 | 4.260 (0.8705)
  BUN Day 9, n= 15: number analyzed (Participants) | 15
  BUN Day 9, n= 15 | 4.263 (0.6977)

46. Secondary Outcome: Period 1: Change From Baseline in Clinical Chemistry Parameter of Alkaline Phosphatase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Lactate Dehydrogenase (LDH), Gamma-glutamyl Transferase (GGT), and Creatine Phosphokinase (CK)
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameter like alkaline phosphatase, ALT, AST, LDH, GGT and CK. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
International units per Liter
  Alkaline phosphatase, Day 7 | -2.6 (5.10)
  Alkaline phosphatase, Day 14 | 2.4 (6.91)
  AST, Day 7 | -6.2 (4.59)
  AST, Day 14 | -6.9 (4.95)
  ALT, Day 7 | -2.1 (7.26)
  ALT, Day 14 | -6.2 (6.98)
  GGT Day 7 | 0.2 (2.32)
  GGT Day 14 | -1.7 (3.63)
  LDH, Day 7 | -14.6 (13.07)
  LDH, Day 14 | -12.0 (16.25)
  CK, Day 7 | -103.0 (127.10)
  CK, Day 14 | -99.2 (135.80)

47. Secondary Outcome: Period 2: Change From Baseline in Clinical Chemistry Parameter of Alkaline Phosphatase, ALT, AST, LDH, GGT, and CK
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of alkaline phosphatase, ALT, AST, LDH, GGT and CK. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
International units per Liter
  Alkaline phosphatase, Day 3, n= 16 | 3.7 (3.48)
  Alkaline phosphatase, Day 7, n= 15: number analyzed (Participants) | 15
  Alkaline phosphatase, Day 7, n= 15 | 2.6 (3.64)
  Alkaline phosphatase, Day 9, n= 15: number analyzed (Participants) | 15
  Alkaline phosphatase, Day 9, n= 15 | -1.0 (3.98)
  AST, Day 3, n= 16 | -1.4 (1.31)
  AST, Day 7, n= 15: number analyzed (Participants) | 15
  AST, Day 7, n= 15 | -0.5 (2.45)
  AST, Day 9, n= 15: number analyzed (Participants) | 15
  AST, Day 9, n= 15 | -0.1 (2.13)
  ALT, Day 3, n= 16 | -2.0 (1.63)
  ALT, Day 7, n= 15: number analyzed (Participants) | 15
  ALT, Day 7, n= 15 | -1.9 (2.76)
  ALT, Day 9, n= 15: number analyzed (Participants) | 15
  ALT, Day 9, n= 15 | -0.7 (4.56)
  GGT, Day 3, n= 16 | -0.9 (1.18)
  GGT, Day 7, n= 15: number analyzed (Participants) | 15
  GGT, Day 7, n= 15 | -1.4 (1.50)
  GGT, Day 9, n= 15: number analyzed (Participants) | 15
  GGT, Day 9, n= 15 | -1.9 (2.55)
  LDH, Day 3, n= 16 | -7.0 (11.98)
  LDH, Day 7, n= 15: number analyzed (Participants) | 15
  LDH, Day 7, n= 15 | -8.2 (12.73)
  LDH, Day 9, n= 15: number analyzed (Participants) | 15
  LDH, Day 9, n= 15 | -7.0 (11.98)
  CK, Day 3, n= 16 | 3.4 (29.12)
  CK, Day 7, n= 15: number analyzed (Participants) | 15
  CK, Day 7, n= 15 | 11.3 (33.83)
  CK, Day 9, n= 15: number analyzed (Participants) | 15
  CK, Day 9, n= 15 | -2.3 (22.65)

48. Secondary Outcome: Period 1: Absolute Values of Clinical Chemistry Parameter of Alkaline Phosphatase, ALT, AST, LDH, GGT, and CK
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of alkaline phosphatase, ALT, AST, LDH, GGT and CK. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
International units per Liter
  Alkaline phosphatase, Baseline | 60.9 (9.33)
  Alkaline phosphatase, Day 7 | 58.3 (8.36)
  Alkaline phosphatase, Day 14 | 63.4 (8.82)
  AST, Baseline | 24.6 (6.16)
  AST, Day 7 | 18.4 (4.79)
  AST, Day 14 | 17.6 (3.46)
  ALT, Baseline | 26.6 (10.44)
  ALT, Day 7 | 24.4 (13.28)
  ALT, Day 14 | 20.4 (8.59)
  GGT Baseline | 1.76 (1.016)
  GGT Day 7 | 1.91 (0.752)
  GGT Day 14 | 2.40 (1.035)
  LDH, Baseline | 138.0 (19.77)
  LDH, Day 7 | 123.4 (19.67)
  LDH, Day 9 | 126.0 (19.50)
  CK, Baseline | 219.6 (150.90)
  CK, Day 7 | 116.6 (49.16)
  CK, Day 14 | 120.4 (62.41)

49. Secondary Outcome: Period 2: Absolute Values of Clinical Chemistry Parameter of Alkaline Phosphatase, ALT, AST, LDH, GGT, and CK
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of alkaline phosphatase, ALT, AST, LDH, GGT and CK. Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
International units per Liter
  Alkaline phosphatase, Baseline Day 3, n= 16 | 63.4 (8.82)
  Alkaline phosphatase, Day 3, n= 16 | 67.1 (10.45)
  Alkaline phosphatase, Day 7, n= 15: number analyzed (Participants) | 15
  Alkaline phosphatase, Day 7, n= 15 | 65.4 (9.81)
  Alkaline phosphatase, Day 9, n= 15: number analyzed (Participants) | 15
  Alkaline phosphatase, Day 9, n= 15 | 61.8 (9.65)
  AST, Baseline, n= 16 | 17.6 (3.46)
  AST, Day 3, n= 16 | 16.2 (3.04)
  AST, Day 7, n= 15: number analyzed (Participants) | 15
  AST, Day 7, n= 15 | 17.2 (3.38)
  AST, Day 9, n= 15: number analyzed (Participants) | 15
  AST, Day 9, n= 15 | 17.6 (3.83)
  ALT, Baseline, n= 16 | 20.4 (8.59)
  ALT, Day 3, n= 16 | 18.4 (7.87)
  ALT, Day 7, n= 15: number analyzed (Participants) | 15
  ALT, Day 7, n= 15 | 18.5 (8.31)
  ALT, Day 9, n= 15: number analyzed (Participants) | 15
  ALT, Day 9, n= 15 | 19.7 (9.43)
  GGT, Baseline, n= 16 | 2.40 (1.035)
  GGT, Day 3, n= 16 | 2.14 (1.065)
  GGT, Day 7, n= 15: number analyzed (Participants) | 15
  GGT, Day 7, n= 15 | 2.41 (0.828)
  GGT, Day 9, n= 15: number analyzed (Participants) | 15
  GGT, Day 9, n= 15 | 1.95 (0.673)
  LDH, Baseline, n= 16 | 126.0 (19.50)
  LDH, Day 3, n= 16 | 119.0 (19.37)
  LDH, Day 7, n= 15: number analyzed (Participants) | 15
  LDH, Day 7, n= 15 | 118.0 (13.93)
  LDH, Day 9, n= 15: number analyzed (Participants) | 15
  LDH, Day 9, n= 15 | 119.2 (17.70)
  CK, Baseline, n= 16 | 120.4 (62.41)
  CK, Day 3, n= 16 | 123.8 (51.53)
  CK, Day 7, n= 15: number analyzed (Participants) | 15
  CK, Day 7, n= 15 | 135.8 (66.33)
  CK, Day 9, n= 15: number analyzed (Participants) | 15
  CK, Day 9, n= 15 | 122.2 (54.94)

50. Secondary Outcome: Period 1: Change From Baseline in Clinical Chemistry Parameter of Lipase and Amylase
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of lipase and amylase. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Units per Liter
  Amylase, Day 7 | -2.3 (9.68)
  Amylase, Day 14 | -2.8 (10.48)
  Lipase, Day 7 | -4.0 (8.93)
  Lipase, Day 14 | -5.3 (12.69)

51. Secondary Outcome: Period 2: Change From Baseline in Clinical Chemistry Parameter of Lipase and Amylase
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of lipase and amylase. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Units per Liter
  Amylase, Day 3, n= 16 | 3.3 (8.93)
  Amylase, Day 7, n= 15: number analyzed (Participants) | 15
  Amylase, Day 7, n= 15 | -1.9 (6.77)
  Amylase, Day 9, n= 15: number analyzed (Participants) | 15
  Amylase, Day 9, n= 15 | 1.1 (6.32)
  Lipase, Day 3, n= 16 | 7.7 (21.62)
  Lipase, Day 7, n= 15: number analyzed (Participants) | 15
  Lipase, Day 7, n= 15 | 0.0 (8.20)
  Lipase, Day 9, n= 15: number analyzed (Participants) | 15
  Lipase, Day 9, n= 15 | 3.5 (3.89)

52. Secondary Outcome: Period 1: Absolute Values of Chemistry Parameters of Lipase and Amylase
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of lipase and amylase. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Units per Liter
  Amylase, Baseline | 56.4 (14.66)
  Amylase, Day 7 | 54.1 (13.15)
  Amylase, Day 14 | 53.6 (14.48)
  Lipase, Baseline | 22.2 (14.00)
  Lipase, Day 7 | 18.2 (9.72)
  Lipase, Day 14 | 16.9 (14.65)

53. Secondary Outcome: Period 2: Absolute Values of Chemistry Parameters of Lipase and Amylase
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of lipase and amylase. Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Units per Liter
  Amylase, Baseline, n= 16 | 53.6 (14.48)
  Amylase, Day 3, n= 16 | 56.8 (19.32)
  Amylase, Day 7, n= 15: number analyzed (Participants) | 15
  Amylase, Day 7, n= 15 | 52.7 (12.97)
  Amylase, Day 9, n= 15: number analyzed (Participants) | 15
  Amylase, Day 9, n= 15 | 55.7 (13.39)
  Lipase, Baseline, n= 16 | 16.9 (14.65)
  Lipase, Day 3, n= 16 | 24.6 (34.82)
  Lipase, Day 7, n= 15: number analyzed (Participants) | 15
  Lipase, Day 7, n= 15 | 17.5 (10.69)
  Lipase, Day 9, n= 15: number analyzed (Participants) | 15
  Lipase, Day 9, n= 15 | 21.0 (14.16)

54. Secondary Outcome: Period 1: Change From Baseline in Clinical Chemistry Parameter of Total Bilirubin, Direct Bilirubin, and Creatinine
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of total bilirubin, direct bilirubin, and creatinine. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Micromoles per liter
  Creatinine, Day 7 | 5.69 (3.508)
  Creatinine, Day 14 | 7.36 (4.833)
  Total bilirubin, Day 7 | 2.25 (4.756)
  Total bilirubin, Day 14 | 2.10 (5.109)
  Direct bilirubin, Day 7 | 0.15 (0.634)
  Direct bilirubin, Day 14 | 0.64 (0.699)

55. Secondary Outcome: Period 2: Change From Baseline in Clinical Chemistry Parameter of Total Bilirubin, Direct Bilirubin, and Creatinine
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of total bilirubin, direct bilirubin, and creatinine. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Micromoles per liter
  Creatinine, Day 3, n= 16 | -2.34 (3.755)
  Creatinine, Day 7, n= 15: number analyzed (Participants) | 15
  Creatinine, Day 7, n= 15 | 3.53 (3.802)
  Creatinine, Day 9, n= 15: number analyzed (Participants) | 15
  Creatinine, Day 9, n= 15 | 0.28 (3.569)
  Total bilirubin, Day 3, n= 16 | -0.82 (3.475)
  Total bilirubin, Day 7, n= 15: number analyzed (Participants) | 15
  Total bilirubin, Day 7, n= 15 | -0.26 (2.466)
  Total bilirubin, Day 9, n= 15: number analyzed (Participants) | 15
  Total bilirubin, Day 9, n= 15 | -1.91 (2.252)
  Direct bilirubin, Day 3, n= 16 | -0.26 (0.534)
  Direct bilirubin, Day 7, n= 15: number analyzed (Participants) | 15
  Direct bilirubin, Day 7, n= 15 | -0.03 (0.547)
  Direct bilirubin, Day 9, n= 15: number analyzed (Participants) | 15
  Direct bilirubin, Day 9, n= 15 | -0.49 (0.501)

56. Secondary Outcome: Period 1: Absolute Values of Clinical Chemistry Parameter of Total Bilirubin, Direct Bilirubin, and Creatinine
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of total bilirubin, direct bilirubin, and creatinine. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Micromoles per liter
  Creatinine, Baseline | 80.16 (10.103)
  Creatinine, Day 7 | 85.85 (9.586)
  Creatinine, Day 14 | 87.52 (10.058)
  Total bilirubin, Baseline | 9.64 (6.143)
  Total bilirubin, Day 7 | 11.89 (6.781)
  Total bilirubin, Day 14 | 11.74 (7.046)
  Direct bilirubin, Baseline | 1.76 (1.016)
  Direct bilirubin, Day 7 | 1.91 (0.752)
  Direct bilirubin, Day 14 | 2.40 (1.035)

57. Secondary Outcome: Period 2: Absolute Values of Clinical Chemistry Parameter of Total Bilirubin, Direct Bilirubin, and Creatinine
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of total bilirubin, direct bilirubin, creatinine and uric acid. Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Micromoles per liter
  Creatinine, Baseline, n= 16 | 87.52 (10.058)
  Creatinine, Day 3, n= 16 | 85.18 (10.314)
  Creatinine, Day 7, n= 15: number analyzed (Participants) | 15
  Creatinine, Day 7, n= 15 | 91.53 (9.504)
  Creatinine, Day 9, n= 15: number analyzed (Participants) | 15
  Creatinine, Day 9, n= 15 | 88.27 (9.916)
  Total bilirubin, Baseline, n= 16 | 11.44 (6.022)
  Total bilirubin, Day 3, n= 16 | 10.62 (7.886)
  Total bilirubin, Day 7, n= 15: number analyzed (Participants) | 15
  Total bilirubin, Day 7, n= 15 | 11.33 (5.487)
  Total bilirubin, Day 9, n= 15: number analyzed (Participants) | 15
  Total bilirubin, Day 9, n= 15 | 9.68 (4.603)
  Direct bilirubin, Baseline, n= 16 | 2.40 (1.035)
  Direct bilirubin, Day 3, n= 16 | 2.14 (1.065)
  Direct bilirubin, Day 7, n= 15: number analyzed (Participants) | 15
  Direct bilirubin, Day 7, n= 15 | 2.41 (0.828)
  Direct bilirubin, Day 9, n= 15: number analyzed (Participants) | 15
  Direct bilirubin, Day 9, n= 15 | 1.95 (0.673)

58. Secondary Outcome: Period 1: Change From Baseline in Clinical Chemistry Parameter of Total Protein, Albumin and Globulin
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of of total protein, albumin and globulin. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Grams per Liter
  Total Protein, Day 7 | 2.6 (3.20)
  Total Protein, Day 14 | 2.9 (2.66)
  Globulin, Day 7 | 2.5 (1.37)
  Globulin, Day 14 | 2.8 (1.91)
  Albumin, Day 7 | 0.1 (2.22)
  Albumin, Day 14 | 0.1 (2.05)

59. Secondary Outcome: Period 2: Change From Baseline in Clinical Chemistry Parameter of Total Protein, Albumin and Globulin
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of total protein, albumin and globulin. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Grams per Liter
  Total Protein, Day 3, n= 16 | 0.1 (2.68)
  Total Protein, Day 7, n= 15: number analyzed (Participants) | 15
  Total Protein, Day 7, n= 15 | 3.1 (2.85)
  Total Protein, Day 9, n= 15: number analyzed (Participants) | 15
  Total Protein, Day 9, n= 15 | 0.8 (3.28)
  Globulin, Day 3, n= 16 | 0.2 (1.17)
  Globulin, Day 7, n= 15: number analyzed (Participants) | 15
  Globulin, Day 7, n= 15 | 2.3 (0.96)
  Globulin, Day 9, n= 15: number analyzed (Participants) | 15
  Globulin, Day 9, n= 15 | 0.2 (1.08)
  Albumin, Day 3, n= 16 | -0.1 (1.95)
  Albumin, Day 7, n= 15: number analyzed (Participants) | 15
  Albumin, Day 7, n= 15 | 0.9 (2.20)
  Albumin, Day 9, n= 15: number analyzed (Participants) | 15
  Albumin, Day 9, n= 15 | 0.6 (2.50)

60. Secondary Outcome: Period 1: Absolute Values of Clinical Chemistry Parameter of Total Protein, Albumin and Globulin
Description: Blood samples were collected at indicated time-points for analysis for clinical chemistry parameter of total protein, albumin and globulin. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Grams per Liter
  Total Protein, Baseline | 69.8 (3.64)
  Total Protein, Day 7 | 72.4 (3.70)
  Total Protein, Day 14 | 72.6 (3.10)
  Globulin, Baseline | 25.9 (2.50)
  Globulin, Day 7 | 28.4 (2.60)
  Globulin, Day 14 | 28.7 (1.99)
  Albumin, Baseline | 43.9 (2.36)
  Albumin, Day 7 | 44.0 (1.90)
  Albumin, Day 14 | 43.9 (2.41)

61. Secondary Outcome: Period 2: Absolute Values of Clinical Chemistry Parameter of Total Protein, Albumin and Globulin
Description: as for outcome 57
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Grams per Liter
  Total Protein, Baseline, n= 16 | 72.6 (3.10)
  Total Protein, Day 3, n= 16 | 72.8 (2.96)
  Total Protein, Day 7, n= 15: number analyzed (Participants) | 15
  Total Protein, Day 7, n= 15 | 75.7 (2.89)
  Total Protein, Day 9, n= 15: number analyzed (Participants) | 15
  Total Protein, Day 9, n= 15 | 73.3 (2.61)
  Globulin, Baseline, n= 16 | 28.7 (1.99)
  Globulin, Day 3, n= 16 | 28.9 (2.31)
  Globulin, Day 7, n= 15: number analyzed (Participants) | 15
  Globulin, Day 7, n= 15 | 30.9 (1.96)
  Globulin, Day 9, n= 15: number analyzed (Participants) | 15
  Globulin, Day 9, n= 15 | 28.8 (1.90)
  Albumin, Baseline, n= 16 | 43.9 (2.41)
  Albumin, Day 3, n= 16 | 43.9 (1.89)
  Albumin, Day 7, n= 15: number analyzed (Participants) | 15
  Albumin, Day 7, n= 15 | 44.8 (2.08)
  Albumin, Day 9, n= 15: number analyzed (Participants) | 15
  Albumin, Day 9, n= 15 | 44.5 (1.73)

62. Secondary Outcome: Period 1: Change From Baseline in Specific Gravity of Urine
Description: Urine samples were collected at indicated time points for the assessment of specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Ratio
  Day 7 | 0.0007 (0.01085)
  Day 14 | 0.0011 (0.00941)

63. Secondary Outcome: Period 2: Change From Baseline in Specific Gravity of Urine
Description: Urine samples were collected at indicated time points for the assessment of specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Ratio
  Day 3, n= 16 | 0.0031 (0.00666)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | 0.0024 (0.00608)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | 0.0005 (0.00872)

64. Secondary Outcome: Period 1: Absolute Values of Specific Gravity of Urine
Description: Urine samples were collected at indicated time points for the assessment of specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Ratio
  Baseline | 1.0136 (0.01095)
  Day 7 | 1.0143 (0.00556)
  Day 14 | 1.0147 (0.00789)

65. Secondary Outcome: Period 2: Absolute Values of Specific Gravity of Urine
Description: Urine samples were collected at indicated time points for the assessment of specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Ratio
  Baseline, n= 16 | 1.0147 (0.00789)
  Day 3, n= 16 | 1.0178 (0.00584)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | 1.0170 (0.00655)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | 1.0151 (0.00788)

66. Secondary Outcome: Period 1: Change From Baseline in Potential of Hydrogen (pH) of Urine
Description: Urine samples were collected at indicated time points for the assessment of Urinary pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
pH
  Day 7 | -0.34 (0.397)
  Day 14 | -0.19 (0.544)

67. Secondary Outcome: Period 2: Change From Baseline in pH of Urine
Description: Urine samples were collected at indicated time points for the assessment of Urinary pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
pH
  Day 3, n= 16 | 0.19 (0.479)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | 0.10 (0.471)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | 0.10 (0.507)

68. Secondary Outcome: Period 1: Absolute Values of pH of Urine
Description: Urine samples were collected at indicated time points for the assessment of Urinary pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
pH
  Baseline | 6.22 (0.446)
  Day 7 | 5.88 (0.289)
  Day 14 | 6.03 (0.531)

69. Secondary Outcome: Period 2: Absolute Values of pH of Urine
Description: Urine samples were collected at indicated time points for the assessment of Urinary pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
pH
  Baseline, n= 16 | 6.03 (0.531)
  Day 3, n= 16 | 6.22 (0.482)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | 6.07 (0.320)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | 6.07 (0.320)

70. Secondary Outcome: Period 1: Change From Baseline in Urine Urobilinogen
Description: Urine samples were collected at indicated time points for the assessment of urine urobilinogen. Baseline was defined as Day -1 for Period 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Micromoles per liter
  Day 7 | -2.5395 (5.45976)
  Day 14 | -2.5395 (5.45976)

71. Secondary Outcome: Period 2: Change From Baseline in Urine Urobilinogen
Description: Urine samples were collected at indicated time points for the assessment of urine urobilinogen. Baseline was defined as Period 1 Day 14 for Period 2. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Micromoles per liter
  Day 3, n= 16 | 0.0000 (0.00000)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | 0.0000 (0.00000)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | 0.0000 (0.00000)

72. Secondary Outcome: Period 1: Absolute Values of Urine Urobilinogen
Description: Urine samples were collected at indicated time points for the assessment of urine urobilinogen. Baseline was defined as Day -1 for Period 1.
Time Frame: Baseline and at Days 7, 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Micromoles per liter
  Baseline | 5.9255 (5.45976)
  Day 7 | 3.3860 (0.0000)
  Day 14 | 3.3860 (0.0000)

73. Secondary Outcome: Period 2: Absolute Values of Urine Urobilinogen
Description: Urine samples were collected at indicated time points for the assessment of urine urobilinogen. Baseline was defined as Period 1 Day 14 for Period 2.
Time Frame: Baseline and at Days 3, 7, 9
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Micromoles per liter
  Baseline, n= 16 | 3.3860 (0.0000)
  Day 3, n= 16 | 3.3860 (0.0000)
  Day 7, n= 15: number analyzed (Participants) | 15
  Day 7, n= 15 | 3.3860 (0.0000)
  Day 9, n= 15: number analyzed (Participants) | 15
  Day 9, n= 15 | 3.3860 (0.0000)

74. Secondary Outcome: Period 1: Change From Baseline in Heart Rate
Description: as for outcome 70
Time Frame: Baseline and at Day 1, 2 and 4 hours post-dose
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Beats per minute
  Day 1, 2 hours post-dose | 1.5 (6.87)
  Day 1, 4 hours post-dose | -3.3 (10.37)

75. Secondary Outcome: Period 2: Change From Baseline in Heart Rate
Description: Twelve-lead ECGs was performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes using an automated ECG machine to measure heart rate. Baseline was defined as Day 1 (Pre-dose) for each Period. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Day 1, 2 and 4 hours post-dose; Day 4, Pre-dose, 2 and 4 hours post-dose; Day 7, Pre-dose, 2 and 4 hours post-dose; Day 9 post-dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Beats per minute
  Day 1, 2 hours post-dose, n= 16 | 5.0 (4.37)
  Day 1, 4 hours post-dose, n= 16 | 2.8 (6.62)
  Day 4, Pre-dose, n= 15: number analyzed (Participants) | 15
  Day 4, Pre-dose, n= 15 | -0.5 (11.10)
  Day 4, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  Day 4, 2 hours post-dose, n= 15 | 3.3 (5.86)
  Day 4, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  Day 4, 4 hours post-dose, n= 15 | -0.3 (5.13)
  Day 7, Pre-dose, n= 15: number analyzed (Participants) | 15
  Day 7, Pre-dose, n= 15 | 0.3 (11.18)
  Day 7, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  Day 7, 2 hours post-dose, n= 15 | 1.8 (6.72)
  Day 7, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  Day 7, 4 hours post-dose, n= 15 | -2.3 (7.08)
  Day 9 post-dose, n= 15: number analyzed (Participants) | 15
  Day 9 post-dose, n= 15 | 2.1 (7.84)

76. Secondary Outcome: Period 1: Absolute Values of Heart Rate
Description: as for outcome 75
Time Frame: Baseline and at Day 1, 2 and 4 hours post-dose
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Beats per minute
  Baseline | 67.6 (8.72)
  Day 1, 2 hours post-dose | 69.1 (11.04)
  Day 1, 4 hours post-dose | 64.4 (11.87)

77. Secondary Outcome: Period 2: Absolute Values of Heart Rate
Description: Twelve-lead ECGs was performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes using an automated ECG machine to measure heart rate. Baseline was defined as Day 1 (Pre-dose) for each Period.
Time Frame: as for outcome 75
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Beats per minute
  Baseline, n= 16 | 66.5 (8.06)
  Day 1, 2 hours post-dose, n= 16 | 71.5 (9.95)
  Day 1, 4 hours post-dose, n= 16 | 69.3 (11.38)
  Day 4, Pre-dose, n= 15: number analyzed (Participants) | 15
  Day 4, Pre-dose, n= 15 | 65.1 (10.48)
  Day 4, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  Day 4, 2 hours post-dose, n= 15 | 68.9 (8.00)
  Day 4, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  Day 4, 4 hours post-dose, n= 15 | 65.3 (8.97)
  Day 7, Pre-dose, n= 15: number analyzed (Participants) | 15
  Day 7, Pre-dose, n= 15 | 65.9 (10.25)
  Day 7, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  Day 7, 2 hours post-dose, n= 15 | 67.4 (6.39)
  Day 7, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  Day 7, 4 hours post-dose, n= 15 | 63.3 (8.31)
  Day 9 post-dose, n= 15: number analyzed (Participants) | 15
  Day 9 post-dose, n= 15 | 67.7 (9.23)

78. Secondary Outcome: Period 1: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval, Fridericia QT Correction Formula (QTcF) Interval, and Bazett QT Correction Formula (QTcB) Interval
Description: Twelve-lead ECGs was performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes using an automated ECG machine to measure PR interval, QRS duration, QT Interal, QTcF Interval and QTcB interval. Baseline was defined as Day 1 (Pre-dose) for each Period. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Day 1, 2 and 4 hours post-dose
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Milliseconds
  PR Interval, Day 1, 2 hours post-dose | 1.5 (9.67)
  PR Interval, Day 1, 4 hours post-dose | -1.9 (8.64)
  QRS Duration, Day 1, 2 hours post-dose | -1.1 (3.68)
  QRS Duration, Day 1, 4 hours post-dose | 0.3 (4.96)
  QT Interval, Day 1, 2 hours post-dose | -7.5 (14.12)
  QT Interval, Day 1, 4 hours post-dose | 5.8 (23.18)
  QTcF Interval, Day 1, 2 hours post-dose | -4.9 (10.63)
  QTcF Interval, Day 1, 4 hours post-dose | -1.3 (10.56)
  QTcB Interval, Day 1, 2 hours post-dose | -4.1 (12.70)
  QTcB Interval, Day 1, 4 hours post-dose | -5.4 (12.39)

79. Secondary Outcome: Period 2: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF Interval, and QTcB Interval
Description: as for outcome 78
Time Frame: as for outcome 75
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Milliseconds
  PR Interval, Day 1, 2 hours post-dose, n= 16 | -6.8 (6.77)
  PR Interval, Day 1, 4 hours post-dose, n= 16 | -3.7 (5.99)
  PR Interval, Day 4, Pre-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 4, Pre-dose, n= 15 | -0.5 (4.56)
  PR Interval, Day 4, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 4, 2 hours post-dose, n= 15 | -6.9 (6.67)
  PR Interval, Day 4, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 4, 4 hours post-dose, n= 15 | -3.9 (7.83)
  PR Interval, Day 7, Pre-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 7, Pre-dose, n= 15 | -2.7 (8.57)
  PR Interval, Day 7, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 7, 2 hours post-dose, n= 15 | -3.3 (7.06)
  PR Interval, Day 7, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 7, 4 hours post-dose, n= 15 | -3.7 (8.53)
  PR Interval, Day 9 post-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 9 post-dose, n= 15 | 1.2 (6.42)
  QRS Duration, Day 1, 2 hours post-dose, n= 16 | -2.5 (4.40)
  QRS Duration, Day 1, 4 hours post-dose, n= 16 | -1.4 (4.69)
  QRS Duration, Day 4, Pre-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 4, Pre-dose, n= 15 | 0.5 (3.44)
  QRS Duration, Day 4, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 4, 2 hours post-dose, n= 15 | 0.5 (5.72)
  QRS Duration, Day 4, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 4, 4 hours post-dose, n= 15 | -0.2 (2.70)
  QRS Duration, Day 7, Pre-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 7, Pre-dose, n= 15 | 3.3 (4.53)
  QRS Duration, Day 7, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 7, 2 hours post-dose, n= 15 | 1.5 (5.15)
  QRS Duration, Day 7, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 7, 4 hours post-dose, n= 15 | 0.3 (3.72)
  QRS Duration, Day 9 post-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 9 post-dose, n= 15 | 3.0 (5.36)
  QT Interval, Day 1, 2 hours post-dose, n= 16 | -12.6 (9.11)
  QT Interval, Day 1, 4 hours post-dose, n= 16 | -1.8 (14.72)
  QT Interval, Day 4, Pre-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 4, Pre-dose, n= 15 | 7.3 (18.27)
  QT Interval, Day 4, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 4, 2 hours post-dose, n= 15 | -6.8 (15.72)
  QT Interval, Day 4, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 4, 4 hours post-dose, n= 15 | 5.6 (14.64)
  QT Interval, Day 7, Pre-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 7, Pre-dose, n= 15 | 3.5 (18.31)
  QT Interval, Day 7, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 7, 2 hours post-dose, n= 15 | -8.4 (16.15)
  QT Interval, Day 7, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 7, 4 hours post-dose, n= 15 | 5.8 (17.37)
  QT Interval, Day 9 post-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 9 post-dose, n= 15 | 4.1 (16.46)
  QTcF Interval, Day 1, 2 hours post-dose, n= 16 | -4.4 (7.29)
  QTcF Interval, Day 1, 4 hours post-dose, n= 16 | 2.4 (7.77)
  QTcF Interval, Day 4, Pre-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 4, Pre-dose, n= 15 | 6.1 (11.17)
  QTcF Interval, Day 4, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 4, 2 hours post-dose, n= 15 | -0.6 (10.91)
  QTcF Interval, Day 4, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 4, 4 hours post-dose, n= 15 | 4.5 (8.22)
  QTcF Interval, Day 7, Pre-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 7, Pre-dose, n= 15 | 4.1 (8.71)
  QTcF Interval, Day 7, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 7, 2 hours post-dose, n= 15 | -5.1 (9.34)
  QTcF Interval, Day 7, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 7, 4 hours post-dose, n= 15 | 0.6 (9.03)
  QTcF Interval, Day 9 post-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 9 post-dose, n= 15 | 7.9 (8.53)
  QTcB Interval, Day 1, 2 hours post-dose, n= 16 | 0.7 (8.83)
  QTcB Interval, Day 1, 4 hours post-dose, n= 16 | 4.7 (8.49)
  QTcB Interval, Day 4, Pre-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 4, Pre-dose, n= 15 | 5.5 (18.50)
  QTcB Interval, Day 4, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 4, 2 hours post-dose, n= 15 | 2.5 (12.37)
  QTcB Interval, Day 4, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 4, 4 hours post-dose, n= 15 | 4.3 (8.52)
  QTcB Interval, Day 7, Pre-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 7, Pre-dose, n= 15 | 4.6 (16.31)
  QTcB Interval, Day 7, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 7, 2 hours post-dose, n= 15 | -3.2 (11.64)
  QTcB Interval, Day 7, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 7, 4 hours post-dose, n= 15 | -1.7 (12.06)
  QTcB Interval, Day 9 post-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 9 post-dose, n= 15 | 10.3 (12.19)

80. Secondary Outcome: Period 1: Absolute Values of ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF Interval, and QTcB Interval
Description: Twelve-lead ECGs was performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes using an automated ECG machine to measure PR interval, QRS duration, QT Interval, QTcF Interval and QTcB interval. Baseline was defined as Day 1 (Pre-dose) for each Period.
Time Frame: Baseline and at Day 1, 2 and 4 hours post-dose
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Milliseconds
  PR Interval, Baseline | 161.3 (16.53)
  PR Interval, Day 1, 2 hours post-dose | 162.8 (19.01)
  PR Interval, Day 1, 4 hours post-dose | 159.4 (19.47)
  QRS Duration, Baseline | 91.0 (8.22)
  QRS Duration, Day 1, 2 hours post-dose | 89.9 (7.54)
  QRS Duration, Day 1, 4 hours post-dose | 91.3 (8.14)
  QT Interval, Baseline | 377.8 (24.84)
  QT Interval, Day 1, 2 hours post-dose | 370.3 (24.74)
  QT Interval, Day 1, 4 hours post-dose | 383.6 (32.12)
  QTcF Interval, Baseline | 391.6 (12.92)
  QTcF Interval, Day 1, 2 hours post-dose | 386.7 (14.33)
  QTcF Interval, Day 1, 4 hours post-dose | 390.3 (18.27)
  QTcB Interval, Baseline | 398.8 (11.28)
  QTcB Interval, Day 1, 2 hours post-dose | 394.6 (15.14)
  QTcB Interval, Day 1, 4 hours post-dose | 393.3 (18.26)

81. Secondary Outcome: Period 2: Absolute Values of ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF Interval, and QTcB Interval
Description: as for outcome 80
Time Frame: as for outcome 75
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Milliseconds
  PR Interval, Baseline, n= 16 | 167.3 (19.46)
  PR Interval, Day 1, 2 hours post-dose, n= 16 | 160.4 (19.73)
  PR Interval, Day 1, 4 hours post-dose, n= 16 | 163.6 (19.04)
  PR Interval, Day 4, Pre-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 4, Pre-dose, n= 15 | 167.1 (22.20)
  PR Interval, Day 4, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 4, 2 hours post-dose, n= 15 | 160.7 (19.59)
  PR Interval, Day 4, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 4, 4 hours post-dose, n= 15 | 163.7 (19.29)
  PR Interval, Day 7, Pre-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 7, Pre-dose, n= 15 | 164.9 (21.11)
  PR Interval, Day 7, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 7, 2 hours post-dose, n= 15 | 164.3 (20.95)
  PR Interval, Day 7, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 7, 4 hours post-dose, n= 15 | 163.9 (22.05)
  PR Interval, Day 9 post-dose, n= 15: number analyzed (Participants) | 15
  PR Interval, Day 9 post-dose, n= 15 | 168.8 (23.70)
  QRS Duration, Baseline, n= 16 | 91.4 (7.87)
  QRS Duration, Day 1, 2 hours post-dose, n= 16 | 88.9 (8.20)
  QRS Duration, Day 1, 4 hours post-dose, n= 16 | 90.1 (7.66)
  QRS Duration, Day 4, Pre-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 4, Pre-dose, n= 15 | 91.8 (8.37)
  QRS Duration, Day 4, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 4, 2 hours post-dose, n= 15 | 91.8 (9.12)
  QRS Duration, Day 4, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 4, 4 hours post-dose, n= 15 | 91.1 (8.51)
  QRS Duration, Day 7, Pre-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 7, Pre-dose, n= 15 | 94.5 (8.25)
  QRS Duration, Day 7, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 7, 2 hours post-dose, n= 15 | 92.7 (7.49)
  QRS Duration, Day 7, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 7, 4 hours post-dose, n= 15 | 91.6 (7.23)
  QRS Duration, Day 9 post-dose, n= 15: number analyzed (Participants) | 15
  QRS Duration, Day 9 post-dose, n= 15 | 94.3 (8.17)
  QT Interval, Baseline, n= 16 | 377.7 (22.66)
  QT Interval, Day 1, 2 hours post-dose, n= 16 | 365.1 (23.71)
  QT Interval, Day 1, 4 hours post-dose, n= 16 | 375.9 (30.14)
  QT Interval, Day 4, Pre-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 4, Pre-dose, n= 15 | 385.6 (26.65)
  QT Interval, Day 4, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 4, 2 hours post-dose, n= 15 | 371.5 (27.31)
  QT Interval, Day 4, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 4, 4 hours post-dose, n= 15 | 383.9 (31.05)
  QT Interval, Day 7, Pre-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 7, Pre-dose, n= 15 | 381.7 (22.25)
  QT Interval, Day 7, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 7, 2 hours post-dose, n= 15 | 369.9 (25.66)
  QT Interval, Day 7, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 7, 4 hours post-dose, n= 15 | 384.1 (30.53)
  QT Interval, Day 9 post-dose, n= 15: number analyzed (Participants) | 15
  QT Interval, Day 9 post-dose, n= 15 | 382.4 (26.55)
  QTcF Interval, Baseline, n= 16 | 390.0 (13.48)
  QTcF Interval, Day 1, 2 hours, n= 16 | 385.6 (15.44)
  QTcF Interval, Day 1, 4 hours post-dose, n= 16 | 392.4 (15.95)
  QTcF Interval, Day 4, Pre-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 4, Pre-dose, n= 15 | 395.0 (21.88)
  QTcF Interval, Day 4, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 4, 2 hours post-dose, n= 15 | 388.3 (17.56)
  QTcF Interval, Day 4, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 4, 4 hours post-dose, n= 15 | 393.4 (18.97)
  QTcF Interval, Day 7, Pre-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 7, Pre-dose, n= 15 | 393.0 (18.42)
  QTcF Interval, Day 7, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 7, 2 hours post-dose, n= 15 | 383.8 (16.19)
  QTcF Interval, Day 7, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 7, 4 hours post-dose, n= 15 | 389.5 (18.06)
  QTcF Interval, Day 9 post-dose, n= 15: number analyzed (Participants) | 15
  QTcF Interval, Day 9 post-dose, n= 15 | 396.8 (18.51)
  QTcB Interval, Baseline, n= 16 | 395.7 (14.19)
  QTcB Interval, Day 1, 2 hours post-dose, n= 16 | 396.4 (17.29)
  QTcB Interval, Day 1, 4 hours post-dose, n= 16 | 400.4 (16.20)
  QTcB Interval, Day 4, Pre-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 4, Pre-dose, n= 15 | 399.2 (25.96)
  QTcB Interval, Day 4, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 4, 2 hours post-dose, n= 15 | 396.2 (16.01)
  QTcB Interval, Day 4, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 4, 4 hours post-dose, n= 15 | 398.0 (17.53)
  QTcB Interval, Day 7, Pre-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 7, Pre-dose, n= 15 | 398.3 (23.83)
  QTcB Interval, Day 7, 2 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 7, 2 hours post-dose, n= 15 | 390.5 (13.31)
  QTcB Interval, Day 7, 4 hours post-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 7, 4 hours post-dose, n= 15 | 391.9 (16.35)
  QTcB Interval, Day 9 post-dose, n= 15: number analyzed (Participants) | 15
  QTcB Interval, Day 9 post-dose, n= 15 | 404.0 (20.62)

82. Secondary Outcome: Period 1: Change From Baseline in Temperature
Description: Temperature was assessed at indicated time-points. Baseline was defined as Day 1 (Pre-dose) for each Period. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4, 5 and 7
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Degree Celsius
  Day 2 | -0.16 (0.400)
  Day 3 | -0.15 (0.576)
  Day 4 | -0.09 (0.406)
  Day 5 | -0.15 (0.371)
  Day 7 | -0.24 (0.491)

83. Secondary Outcome: Period 2: Change From Baseline in Temperature
Description: as for outcome 82
Time Frame: Baseline and at Days 4, 7, 9, and 10
Population: Safety Population. Only those participants with data available at the specified time points
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Degree Celsius
  Day 4 | -0.10 (0.344)
  Day 7 | -0.07 (0.337)
  Day 9 | -0.01 (0.386)
  Day 10 | 0.07 (0.320)

84. Secondary Outcome: Period 1: Absolute Values of Temperature
Description: Temperature was assessed at indicated time-points. Baseline was defined as Day 1 (Pre-dose) for each Period.
Time Frame: Baseline and at Days 2, 3, 4, 5 and 7
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Degree Celsius
  Baseline | 36.49 (0.298)
  Day 2 | 36.33 (0.342)
  Day 3 | 36.34 (0.456)
  Day 4 | 36.41 (0.431)
  Day 5 | 36.34 (0.360)
  Day 7 | 36.25 (0.407)

85. Secondary Outcome: Period 2: Absolute Values of Temperature
Description: Temperature was assessed at indicated time-points. Baseline was defined as Day 1 (Pre-dose) for each Period.
Time Frame: Baseline and at Days 4, 7, 9, and 10
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Degree Celsius
  Baseline, n= 16 | 36.49 (0.257)
  Day 4, n=15: number analyzed (Participants) | 15
  Day 4, n=15 | 36.37 (0.348)
  Day 7, n=15: number analyzed (Participants) | 15
  Day 7, n=15 | 36.40 (0.421)
  Day 9, n=15: number analyzed (Participants) | 15
  Day 9, n=15 | 36.46 (0.378)
  Day 10, n=15: number analyzed (Participants) | 15
  Day 10, n=15 | 36.53 (0.282)

86. Secondary Outcome: Period 1: Change From Baseline in Pulse Rate
Description: Pulse rate was assessed in the semi-recumbent position with a completely automated device at indicated time-points. Baseline was defined as Day 1 (Pre-dose) for each Period. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4, 5 and 7
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Beats per minute
  Day 2 | -1.2 (9.77)
  Day 3 | -3.8 (9.94)
  Day 4 | -4.0 (9.67)
  Day 5 | -1.6 (10.47)
  Day 7 | -7.6 (7.83)

87. Secondary Outcome: Period 2: Change From Baseline in Pulse Rate
Description: as for outcome 86
Time Frame: Baseline and at Days 4, 7, 9, and 10
Population: Safety Population. Only those participants with data available at the specified time points
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Beats per minute
  Day 4 | 2.4 (18.62)
  Day 7 | 1.9 (15.62)
  Day 9 | -0.3 (10.20)
  Day 10 | 9.5 (11.12)

88. Secondary Outcome: Period 1: Absolute Values of Pulse Rate
Description: Pulse rate was assessed in the semi-recumbent position with a completely automated device at indicated time-points. Baseline was defined as Day 1 (Pre-dose) for each Period.
Time Frame: Baseline and at Days 2, 3, 4, 5 and 7
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Beats per minute
  Baseline | 73.9 (9.24)
  Day 2 | 72.8 (10.14)
  Day 3 | 70.1 (11.18)
  Day 4 | 69.9 (10.81)
  Day 5 | 72.3 (12.38)
  Day 7 | 66.3 (10.20)

89. Secondary Outcome: Period 2: Absolute Values of Pulse Rate
Description: as for outcome 88
Time Frame: Baseline and at Days 4, 7, 9, and 10
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Beats per minute
  Baseline, n= 16 | 70.5 (11.33)
  Day 4, n=15: number analyzed (Participants) | 15
  Day 4, n=15 | 71.9 (18.39)
  Day 7, n=15: number analyzed (Participants) | 15
  Day 7, n=15 | 71.4 (14.73)
  Day 9, n=15: number analyzed (Participants) | 15
  Day 9, n=15 | 69.2 (10.73)
  Day 10, n=15: number analyzed (Participants) | 15
  Day 10, n=15 | 79.0 (12.45)

90. Secondary Outcome: Period 1: Change From Baseline in Respiratory Rate
Description: Respiratory rate was assessed at indicated time-points. Baseline was defined as Day 1 (Pre-dose) for each Period. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4, 5 and 7
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Breaths per minute
  Day 2 | -1.5 (2.00)
  Day 3 | -0.5 (3.14)
  Day 4 | -0.5 (2.37)
  Day 5 | 1.3 (2.52)
  Day 7 | 0.6 (3.24)

91. Secondary Outcome: Period 2: Change From Baseline in Respiratory Rate
Description: as for outcome 90
Time Frame: Baseline and at Days 4, 7, 9, and 10
Population: Safety Population. Only those participants with data available at the specified time points
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Breaths per minute
  Day 4 | -3.2 (3.61)
  Day 7 | -2.4 (2.85)
  Day 9 | -0.8 (2.11)
  Day 10 | -1.5 (2.33)

92. Secondary Outcome: Period 1: Absolute Values of Respiratory Rate
Description: Respiratory rate was assessed at indicated time-points. Baseline was defined as Day 1 (Pre-dose) for each Period.
Time Frame: Baseline and at Days 2, 3, 4, 5 and 7
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Breaths per minute
  Baseline | 14.0 (1.63)
  Day 2 | 12.5 (1.37)
  Day 3 | 13.5 (2.48)
  Day 4 | 13.5 (2.00)
  Day 5 | 15.3 (2.05)
  Day 7 | 14.6 (2.70)

93. Secondary Outcome: Period 2: Absolute Values of Respiratory Rate
Description: Respiratory rate was assessed at indicated time-points. Baseline was defined as Day 1 (Pre-dose) for each Period.
Time Frame: Baseline and at Days 4, 7, 9, and 10
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Breaths per minute
  Baseline, n= 16 | 15.6 (2.22)
  Day 4, n=15: number analyzed (Participants) | 15
  Day 4, n=15 | 12.5 (2.67)
  Day 7, n=15: number analyzed (Participants) | 15
  Day 7, n=15 | 13.3 (2.35)
  Day 9, n=15: number analyzed (Participants) | 15
  Day 9, n=15 | 14.9 (1.49)
  Day 10, n=15: number analyzed (Participants) | 15
  Day 10, n=15 | 14.3 (1.49)

94. Secondary Outcome: Period 1: Change From Baseline in Blood Pressure
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) was assessed in the semi-recumbent position with a completely automated device at indicated time-points. Baseline was defined as Day 1 (Pre-dose) for each Period. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 2, 3, 4, 5 and 7
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Millimeters of mercury
  SBP, Day 2 | 1.4 (8.96)
  SBP, Day 3 | -1.8 (8.54)
  SBP, Day 4 | -2.7 (6.16)
  SBP, Day 5 | -2.3 (8.81)
  SBP, Day 7 | 0.8 (9.47)
  DBP, Day 2 | 0.1 (8.33)
  DBP, Day 3 | -1.6 (7.20)
  DBP, Day 4 | 0.1 (7.89)
  DBP, Day 5 | -1.4 (6.20)
  DBP, Day 7 | 2.9 (7.58)

95. Secondary Outcome: Period 2: Change From Baseline in Blood Pressure
Description: SBP and DBP was assessed in the semi-recumbent position with a completely automated device at indicated time-points. Baseline was defined as Day 1 (Pre-dose) for each Period. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and at Days 4, 7, 9, and 10
Population: Safety Population. Only those participants with data available at the specified time points
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Millimeters of mercury
  SBP, Day 4 | -0.3 (5.07)
  SBP, Day 7 | 1.1 (8.95)
  SBP, Day 9 | -1.7 (6.91)
  SBP, Day 10 | 4.1 (7.79)
  DBP, Day 4 | 0.1 (4.96)
  DBP, Day 7 | 3.7 (5.70)
  DBP, Day 9 | -4.0 (5.26)
  DBP, Day 10 | -2.1 (8.18)

96. Secondary Outcome: Period 1: Absolute Values of Blood Pressure
Description: SBP and DBP was assessed in the semi-recumbent position with a completely automated device at indicated time-points. Baseline was defined as Day 1 (Pre-dose) for each Period.
Time Frame: Baseline and at Days 2, 3, 4, 5 and 7
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Millimeters of mercury
  SBP, Baseline | 123.3 (8.27)
  SBP, Day 2 | 124.7 (9.60)
  SBP, Day 3 | 121.5 (7.70)
  SBP, Day 4 | 120.6 (8.47)
  SBP, Day 5 | 121.0 (6.95)
  SBP, Day 7 | 124.1 (10.56)
  DBP, Baseline | 75.3 (5.22)
  DBP, Day 2 | 75.4 (9.08)
  DBP, Day 3 | 73.8 (5.69)
  DBP, Day 4 | 75.4 (10.42)
  DBP, Day 5 | 73.9 (5.46)
  DBP, Day 7 | 78.2 (7.57)

97. Secondary Outcome: Period 2: Absolute Values of Blood Pressure
Description: as for outcome 96
Time Frame: Baseline and at Days 4, 7, 9, and 10
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 16
Millimeters of mercury
  SBP, Baseline, n= 16 | 120.4 (7.27)
  SBP, Day 4, n=15: number analyzed (Participants) | 15
  SBP, Day 4, n=15 | 119.3 (7.03)
  SBP, Day 7, n=15: number analyzed (Participants) | 15
  SBP, Day 7, n=15 | 120.8 (10.58)
  SBP, Day 9, n=15: number analyzed (Participants) | 15
  SBP, Day 9, n=15 | 117.9 (7.42)
  SBP, Day 10, n=15: number analyzed (Participants) | 15
  SBP, Day 10, n=15 | 123.7 (8.52)
  DBP, Baseline, n= 16 | 74.4 (6.14)
  DBP, Day 4, n= 15: number analyzed (Participants) | 15
  DBP, Day 4, n= 15 | 74.3 (5.16)
  DBP, Day 7, n= 15: number analyzed (Participants) | 15
  DBP, Day 7, n= 15 | 77.9 (8.98)
  DBP, Day 9, n= 15: number analyzed (Participants) | 15
  DBP, Day 9, n= 15 | 70.3 (7.36)
  DBP, Day 10, n= 15: number analyzed (Participants) | 15
  DBP, Day 10, n= 15 | 72.1 (6.41)

98. Secondary Outcome: Period 2: AUC (0-tau) of GSK3640254
Description: as for outcome 2
Time Frame: Pre-dose, 1 and 2hours, 2 hours 30 minutes, 3 and 3 hour 30 minutes, 4 and 4 hour 30 minutes, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Hours*nanogram per milliliter | 24.53 (26.5)

99. Secondary Outcome: Period 2: Cmax of GSK3640254
Description: as for outcome 3
Time Frame: as for outcome 98
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Nanogram per milliliter | 1.411 (26.4)

100. Secondary Outcome: Period 2: Ctau of GSK3640254
Description: as for outcome 9
Time Frame: Pre-dose, 1 and 2 hours, 2 hours 30 minutes, 3 and 3 hour 30 minutes, 4 and 4 hour 30 minutes, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Nanogram per milliliter | 0.7883 (30.3)

101. Secondary Outcome: Period 2: Time of Maximum Observed Concentration (Tmax) of GSK3640254
Description: Blood samples were collected at indicated time-points for analysis of Tmax. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 98
Population: PK Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Hours | 5.000 [2.50 to 8.00]

102. Secondary Outcome: Period 1: Tmax of TAF
Description: as for outcome 101
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 1 Day 14
Population: PK Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Hours | 1.00 [0.50 to 2.00]

103. Secondary Outcome: Period 2: Tmax of TAF
Description: as for outcome 101
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Hours | 1.000 [0.50 to 2.00]

104. Secondary Outcome: Period 1: Tmax of FTC
Description: as for outcome 101
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 1 Day 14
Population: PK Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Hours | 1.500 [1.00 to 3.00]

105. Secondary Outcome: Period 2: Tmax of FTC
Description: as for outcome 101
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Hours | 1.500 [1.00 to 3.08]

106. Secondary Outcome: Period 1: Tmax of TFV
Description: as for outcome 101
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 1 Day 14
Population: PK Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | TAF/FTC
Number analyzed (Participants) | 16
Hours | 3.000 [1.50 to 4.00]

107. Secondary Outcome: Period 2: Tmax of TFV
Description: as for outcome 101
Time Frame: Pre-dose, 15, 30, 45 minutes, 1 hour, 1 hour 30 minutes, 2, 3, 4, 5, 6, 8, 12 and 24 hours in Period 2 Day 7
Population: PK Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | TAF/FTC+GSK3640254
Number analyzed (Participants) | 15
Hours | 3.000 [1.00 to 5.00]

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected from the start of the study treatment up to Day 24
Description: Non-serious AEs and SAEs were reported for the safety population which comprised of all participants who received at least one dose of study medication.
Arm/Group | TAF/FTC | TAF/FTC+GSK3640254
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 9/16 | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAF/FTC (N=16) | TAF/FTC+GSK3640254 (N=16)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Rash pustular (Infections and infestations) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT03836729/SAP_000.pdf
  • Study Protocol (2018-12-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT03836729/Prot_001.pdf